CLINICAL TRIAL: NCT07340736
Title: Sensory Mechanisms of Manual Dexterity Recovery After Stroke: a Prospective Cohort Study of Prediction and Cerebral Correlates
Acronym: HapticS 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-A00115-44
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Upper Extremity Paresis; Manual Dexterity; Sensory Integration Dysfunction; Vibration
Keywords: stroke; haptic; vibration; sensorimotor impairment; manual dexterity; prediction of recovery; MRI
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke patients in the early subacute phase (Experimental): Patients will be followed for 6 months over three visits. They will undergo validated sensory, motor, and cognitive clinical assessments, as well as MRI scans and manual dexterity tests performed with and without the addition of vibratory stimulation to the fingers, using a tool previously developed as part of this project.
  Interventions: Device: Haptic stimulation device; Other: Brain MRI
- Healthy controls matched in age, sex and laterality with stroke patients (Active Comparator): Healthy control participants will be assessed during a single visit. They will undergo motor, sensory, and cognitive clinical assessments, as well as manual dexterity tasks performed with and without the addition of finger vibrations using a previously developed tool. They will also undergo anatomical, resting-state functional, and diffusion brain MRI sequences. Each healthy participant will be matched to a patient in terms of age, sex, and handedness of the affected limb. For example, if we include a 60-year-old male post-stroke patient who is right-handed and has a right upper-limb impairment, we will include a healthy male participant aged 60 ± 5 years who is also right-handed.
  Interventions: Device: Haptic stimulation device; Other: Brain MRI

INTERVENTIONS:
Device: Haptic stimulation device — Both patients and healthy participants will perform manual dexterity tasks using the Dextrain Manipulandum. In addition, they will receive finger vibrations delivered via rings that we have previously developed. These vibrations will have a frequency of 150 Hz and will be delivered for a duration of 150 ms.
Other: Brain MRI — Subjects and patients will undergo anatomical, resting-state functional, and diffusion brain MRI sequences.

SUMMARY:
In the proposed research, we will assess motor and sensory functions of the hand using clinical tests and a tool designed to measure manual dexterity combined with vibrotactile stimulation. We will also evaluate the integrity of brain structure and function using MRI.

DETAILED DESCRIPTION:
In this study, 90 post-stroke patients will be followed over three visits at 3 weeks, 3 months, and 6 months after stroke. Manual dexterity will be assessed using the Dextrain Manipulandum, both with and without the addition of finger vibrations. These vibrations will be delivered using vibratory rings, a tool that has been developed and is currently being validated in healthy participants and in patients with chronic post-stroke conditions. These measurements will allow us to quantify haptic facilitation, that is the impact of adding finger vibrations on hand motor function.

During each of the three visits, we will also administer validated sensory, motor, and cognitive clinical assessments, as well as anatomical, resting-state functional, and diffusion MRI sequences to investigate brain structure and function in relation to this haptic facilitation. These longitudinal measurements will enable the development of biomarkers of motor recovery of manual dexterity after stroke, with the primary objective of improving the prediction of dexterity recovery using a regression model.

ELIGIBILITY:
Inclusion Criteria:

* First symptomatic stroke, ischaemic or haemorrhagic in the early subacute phase (up to 3 weeks post-stroke)
* Upper limb paresis (≤4/5 MRC Scale)
* Ability to grasp, lift and put down 1 block (from the BBT test)
* Be affiliated to a social security

Exclusion Criteria:

* Presence of another neurological or musculoskeletal condition affecting upper limb movement
* Severe cognitive impairment and/or aphasia with inability to understand and carry out instructions
* Contraindications to MRI (claustrophobia, presence of cochlear implants and/or pacemakers)
* Persons subject to legal protection measures
* Persons subject to judicial protection measures
* Pregnancy
* Life-threatening conditions or conditions requiring follow-up at 6 months
* Epilepsy
* Known hypersensitivity or allergy to silicone

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Gain in the prediction of manual dexterity recovery | 3 months post enrollment
  The primary outcome measure is a 10% improvement in the prediction of the Box and Block Test (BBT) score at 3 and 6 months post-stroke achieved by adding the haptic effect to a multivariate model.

SECONDARY OUTCOMES:
Change in the prediction of the Box and Block Test (BBT) score when taking into account the haptic effect during an index finger force control task. | 3 and 6 months post enrollment
  Determine whether the haptic effect calculated during an index finger force control exercise (using the dextrain manipulandum) measured in the acute phase after stroke can improve the prediction of manual dexterity recovery (Box and Blocks Test, BBT) at 3 months and 6 months after stroke.
Predicting recovery in various clinical tests of motor and sensory function and activity limitations at 3 months and 6 months post-stroke. | 3 and 6 months post enrollment
  Determine whether the haptic effect VS absence of haptic effect improves the prediction of recovery from motor impairment (Fugl Mayer Assessment for Upper Extremity FMA-UE, Purdue Pegboard Test), sensitivity (monofilaments and Nottingham Sensory Assessment), and activity limitations (Stroke Impact Scale) of the upper limb from 3 weeks to 3 and 6 months post-stroke.
Difference in functional and structural connectivity between subgroups with vs without haptic effect at 3 and 6 months | 3 and 6 months post enrollement
  Investigate whether connectivity of fronto-parietal networks at 3 weeks post-stroke predicts recovery of haptic effect and dexterity at 3 and 6 months.
Changes in the structural and functional connectivity of fronto-parietal networks between 3 weeks and 6 months post-stroke | 3 and 6 months post stroke
  A difference in the change in connectivity between subgroups with versus without haptic effect at 6 months will be investigated.
Difference in brain connectivity between brain images of healthy subjects and patients 3 weeks post-stroke and healthy subjects and patients 6 months post-stroke. | 6 months post enrollement
  Compare brain connectivity between the group of healthy subjects and the group of patients at 3 weeks and 6 months post-stroke.
Correlation between the location of the lesion at 3 weeks and the haptic effect and the results of clinical tests | 3 and 6 months post stroke
  These correlations will be done using Voxel Based Lesion Symptoms Mapping technique (VLSM)

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Psychiatrie et Neurosciences, Paris, France

IPD SHARING:
Plan to Share IPD: No